CLINICAL TRIAL: NCT05053763
Title: The 90% Effective Dose of Remimazolam for Duodenoscopy Insertion During ERCP
Brief Title: The 90% Effective Dose of Remimazolam for Duodenoscopy Insertion During ERCP With Alfentanil 10µg/kg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jianbo Yu (Other)
Responsible Party: Sponsor-Investigator, Jianbo Yu, Director, Tianjin Nankai Hospital
Organization: Tianjin Nankai Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TianjinNK RM-ED90
Record Dates: First submitted 2021-09-21; First posted 2021-09-22 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Anesthesia
Keywords: ERCP; remimazolam; alfentanil; ED90
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: age<65 group (Other): The 90% effective dose of remimazolam for duodenoscopy insertion with alfentanil 10µg/kg
  Interventions: Drug: Remimazolam
- Active Comparator:age ≥65 group (Other): The 90% effective dose of remimazolam for duodenoscopy insertion with alfentanil 10µg/kg
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — The study was carried out using a biased coin design up-and-down sequential method, where the dose of remimazolam administered to each patient depended on the response of the previous one with success/failure duodenoscopy insertion during ERCP are required for reliable estimates. The first patient was tested at 0.2mg/kg remimazolam (0.025mg/kg as a step size). Duodenoscopy insertion was conducted when MOAA/S≤1.The response of the patients to the duodenoscopy insertion during ERCP was categorized as either 'success (no movement)' or 'failure (movement). if a patient had a failure duodenoscopy insertion, the dose of remimazolam was increased by 0.025mg/kg in the next subject. If a patient had a successful duodenoscopy insertion the next subject was randomised to receive either a lower dose (with a decrement of 0.025mg/kg), with a probability of b = 0.11, or the same dose, with a probability of 1-b = 0.89.

SUMMARY:
Remimazolam has shown promising results for sedation in colonoscopy . Alfentanil is widely used in the analgesia of ERCP . The purpose of the study was to determine the 90% Effective Dose of Remimazolam for Duodenoscopy Insertion During ERCP With Alfentanil 10µg/kg

DETAILED DESCRIPTION:
1. Title:The 90% Effective Dose of Remimazolam for Duodenoscopy Insertion During ERCP With Alfentanil 10µg/kg 2. Research center: Single center. 3. The population of the study: Age is between 18 and 85 years; ASA I-III levels; Patients undergone elective ERCP surgery, non-intubation patients; 4. Sample size:The sample size was decided based on that of prior Literature.The study was carried out using a biased coin design up-and-down sequential method, where the dose of remimazolam administered to each patient depended on the response of the previous one with success/failure duodenoscopy insertion during ERCP are required for reliable estimates. The first patient recruited received a dose of 0.2mg/kg, based on our past experience.Subsequently, if a patient had a failure duodenoscopy insertion, the dose of remimazolam was increased by 0.025mg/kg in the next subject. If a patient had a successful duodenoscopy insertion the next subject was randomised to receive either a lower dose (with a decrement of 0.025mg/kg), with a probability of b = 0.11, or the same dose, with a probability of 1-b = 0.89.

We defined duodenoscopy insertion a failure was as gross purposeful muscular movement, coughing or vomiting occurring during or within 2 minutes of insertion of duodenoscopy. If BIS>75 and MOAA/S > 1 when 3 min after the intravenous injection of remimazolam, it was considered a failure, and the patient received rescue sedation. Success was depicted when the reactions mentioned earlier were absent.

ELIGIBILITY:
Inclusion Criteria:

* Age is between 18 and 85 years
* ASA I-III levels;
* Patients undergone elective ERCP surgery, non-intubation patients;

Exclusion Criteria:

* Chronic pain with long-term use of analgesics, psychotropic substances (including opioids, NSAIDs, sedatives, antidepressants), alcohol abusers, with known drug allergy;
* BMI<18 or BMI>30;
* Previous abnormal surgical anesthesia recovery history;
* Hypertension or systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 95 mmHg when the patient admission to the operating room
* Suffering from esophageal reflux; • Sedatives, analgesics and antipruritic drugs were used 24 hours before operation;
* Expected difficult intubation ;
* Opioids allergy history;
* Take monoamine oxidase inhibitor or antidepressant within 15 days;
* Pregnant or parturient women;
* Involved in other drug trials within three months;
* Patients who can not communicate well with the researcher

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-12-25 (Estimated); Study Completion 2022-12-25 (Estimated)

PRIMARY OUTCOMES:
The number of success duodenoscopy insertion | 1 day
  success duodenoscopy insertion is defined by no body movement

SECONDARY OUTCOMES:
The number of the occurrence of hypotension | 1 day
  hypotension is defined MAP decrease by 20%
The number of the occurrence of bradycardia | 1 day
  bradycardia is defined lower than 50 beats / min
The number of the occurrence of injection pain | 1 day
  injection pain is defined the patient complained of vascular pain

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Nankai Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Guo Y, Dong SA, Shi J, Chen HR, Liu SS, Wu LL, Wang JH, Zhang L, Li HX, Yu JB. The 90% effective dose (ED90) of remimazolam for inhibiting responses to the insertion of a duodenoscope during ERCP. BMC Anesthesiol. 2024 May 14;24(1):174. doi: 10.1186/s12871-024-02554-1. PMID 38745175